CLINICAL TRIAL: NCT05811637
Title: Istanbul University, Faculty of Health Science, Division of Physiotherapy and Rehabilitation
Brief Title: Investigation of the Effect of Pilates Exercises on Patellofemoral Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Derya Celik, Prof., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D2023
Record Dates: First submitted 2023-03-31; First posted 2023-04-13 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Patellofemoral Pain
Keywords: Patellofemoral pain; core; quality of life; exercise; strength; pilates
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity | interventions — Exercise Movement Techniques

STUDY DESIGN:
Intervention Model Description: Randomized and trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Supervised Rehabilitation (Active Comparator): The supervised rehabilitation focused mainly on strengthening the hip-knee muscles and flexibility exercises for the gastrocnemius and hamstring muscles. Hip and knee targeted strengthening and stretching exercises will be applied for 6 weeks, two sessions a week 12 sessions of all exercises, 3 sets, and 10-15 repetitions of each set.
  Interventions: Other: Supervised Rehabilitation
- Pilates Exercise (Active Comparator): The principles of Pilates exercises will be taught to the patients in the first session, and the evaluation will be made. The exercises, including basic training exercises in the first week, will be performed for 6 weeks, each session lasting 45 minutes, two days a week, each exercise for 8-12 repetitions. The Pilates exercises, consisting of gradually increasing strengthening will be applied under the supervision of a physiotherapist.
  Interventions: Other: Pilates Exercise

INTERVENTIONS:
Other: Pilates Exercise — The program will be applied with the Pilates exercises every week. All patients were evaluated before and after the treatment (6 weeks).
  Arms: Pilates Exercise
Other: Supervised Rehabilitation — The program will be applied with the progression of the supervised rehabilitation in the 4th week
  Arms: Supervised Rehabilitation

SUMMARY:
This study aimed to investigate the effectiveness of Pilates exercises in Patellofemoral pain patients compared to hip and knee combined exercises in improving pain, muscle strength, flexibility, function and quality of life in short term.

DETAILED DESCRIPTION:
Patellofemoral pain is a common condition characterized by pain in anterior knee, around the kneecap. It is known that exercise is beneficial in rehabilitation in general. Exercise programs applied to patients with PFP should include hip and knee-targeted combined exercises. Nowadays, Pilates is used as an effective rehabilitation tool for individuals with musculoskeletal problems, especially in reducing pain and improving function. Therefore, we believe that Pilates exercises can be effective in PFP Considering that PFP is a chronic condition and exercise therapy is one of the main strategies in the treatment. Pilates may be preferred as one of the alternative treatment method.

This randomized controlled study was designed to compare the effects of two different treatment protocols, Group-I (Supervised Rehabilitation) and Group-II (Pilates Exercises). Patients who applied to the Istanbul Physical Therapy and Rehabilitation Training and Research Hospital, Sports Medicine outpatient clinic and were diagnosed with PFP by a specialist physician based on the patient histories, physical examinations, and diagnostic imaging. The estimated desired sample size was at least 14 participants per group. We anticipated a dropout rate of 20%. Therefore, 34 participants were required for each group (Supervised Rehabilitation n=17, Pilates Exercises n=17) of both sexes, ages ranging from 18-45 years. A computer generated randomization list was used to divide the patients into two groups (https://www.randomizer.org/). An 'Informed Consent Form' was obtained from patients by explaining the purpose of the study, the duration of the study, the treatments to be applied, and possible side effects.

ELIGIBILITY:
Inclusion Criteria:

* Having characteristic signs of PFP (retropatellar or peripatellar pain)
* Presence of at least 3 points of retropatellar or peripatellar pain on the Numbered Pain Rating Scale (NPRS) with squatting, climbing stairs, prolonged sitting, or functional activity that burdens the PFP
* Presence of any of the criteria such as tenderness, small effusion in the patellar facet palpation

Exclusion Criteria:

* Patellofemoral dislocation, subluxation, intra-articular knee pathology
* Previous lower extremity surgery, and knee-related trauma
* A history of hip pathology or neurological disorders
* Knee trauma in the last 1 month

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2023-04-15 (Actual); Primary Completion 2023-10-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Functional assessment | 6 weeks
  Kujala Anterior Knee Pain Scale is used to assess the functional disability levels of the patients.
Pain assessment | 6 weeks
  The numerical NPRS is used to measure and monitor the severity of pain. The patients will be asked to rate the severity of the current pain level between 0 and 10 (0 being "no pain" and 10 being the "worst imaginable pain").

SECONDARY OUTCOMES:
Muscle strength assessment | 6 weeks
  Quadriceps strength will be measured using the Lafayette Manual Muscle Tester (Lafayette Instrument-model 01165, USA) handheld dynamometer.
Muscle flexibility assessment | 6 weeks
  The flexibility of the hamstring muscles' length will be measured with the "Sit and Reach Test".
Quality of life assessment | 6 weeks
  The short form SF-36v2 will be used to assess the quality of life. The scale, designed to assess the quality of life, covers physical, social, and psychological conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No